CLINICAL TRIAL: NCT06915246
Title: A Randomized Phase 2 Study of Carmustine Formulated With and Without Ethanol as Part of BEAM Chemotherapy Conditioning for Subjects With Lymphoma Undergoing Autologous Hematopoietic Cell Transplantation (AHCT)
Brief Title: A Study of Carmustine With and Without Ethanol in Subjects With Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VIVUS LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LY-201
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Lymphoma; Non-Hodgkin Lymphoma; Hodgkin Lymphoma
Keywords: Lymphoma; AHCT; BiCNU; Carmustine
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin; Hodgkin Disease | interventions — Carmustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VI-0609 (Experimental): VI-0609 (Carmustine with Propylene Glycol)
  Interventions: Drug: VI-0609
- BiCNU (Active Comparator): BiCNU (Carmustine with Ethanol)
  Interventions: Drug: BiCNU

INTERVENTIONS:
Drug: VI-0609 — Carmustine with Propylene Glycol
  Arms: VI-0609
Drug: BiCNU — Carmustine with Ethanol
  Arms: BiCNU

SUMMARY:
A phase 2 multicenter study of VI-0609 vs BiCNU in the BEAM high-intensity conditioning regimen for AHCT in subjects with lymphomas.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults ≥ 18 years of age with a life expectancy ≥ 6 months;
* Karnofsky performance status ≥ 70%;
* Histologically confirmed Hodgkin lymphoma or Non-Hodgkin lymphoma;
* Candidate for AHCT consolidation therapy as assessed by their treating physician;
* Achieved a complete or partial response;
* Completed collection of at least 2.0 x 10^6 CD34 cells/kg of autologous hematopoietic progenitor cells (HPCs) by apheresis;
* Recovery from non-hematologic toxicities of salvage cytoreductive chemotherapy to ≤ grade 2;
* Clinical laboratory and organ function criteria meeting study ranges/limits LVEF ≥ 50%; FEV1 > 65% of predicted measurement, DLCO ≥ 50% of predicted;
* Seronegative for HIV Ag/Ab combo, HCV, active HBV, and syphilis

Exclusion Criteria:

* Prior high-dose chemotherapy with autologous stem cell transplant, or prior allogeneic transplantation;
* Significant prior external beam dose-limiting radiation to a critical organ based on review of the prior radiation treatment records;
* Use of any other investigational medication or device, or concurrent biological, chemotherapy, or radiation therapy;
* Myelodysplasia or any active malignancy other than HL or NHL, or < 5 years remission from any other prior malignancy;
* Any cytogenetic abnormality in the bone marrow that is known to be associated with or predictive of myelodysplasia;
* Persistent marrow involvement (>10%) with HL or NHL after salvage cytoreductive therapy and before stem cell mobilization;
* Not having sufficient bone marrow harvest to reach adequate cell dose for transplant;
* Active hepatitis B or C viral infection or HBsAg positive;
* Positive HIV antibody;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of infusion-related toxicities | Within 24 hours post infusion
Evaluation of unacceptable toxicities | From start of BEAM through Day 30 post-AHCT

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - City of Hope Phoenix, Goodyear, Arizona
  - City of Hope National Medical Center, Duarte, California
  - City of Hope Atlanta, Newnan, Georgia
  - City of Hope Chicago, Zion, Illinois

IPD SHARING:
Plan to Share IPD: No